CLINICAL TRIAL: NCT01946334
Title: Does Body Position Influence Pressure Recording by High-resolution Manometry ?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-A00507-38; 2013-13 (Other: AP HM)
Record Dates: First submitted 2013-09-11; First posted 2013-09-19 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Anal Incontinence or Constipation
MeSH Terms: conditions — Encopresis; Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients (Experimental)
  Interventions: Device: anorectal manometry and high-resolution three-dimensional

INTERVENTIONS:
Device: anorectal manometry and high-resolution three-dimensional

SUMMARY:
The anorectal manometry is the gold standard in the evaluation of anorectal function.

Several techniques are currently used (balloons, perfused catheters) and are always performed in the supine position.

Few studies have reported the evaluation of sphincter function in the upright position, whereas symptoms of fecal incontinence occur in this position.

Recently developed, high-resolution manometry, thanks to its many mechanical sensors, allows topographic analysis and evaluation of anorectal function more acurate. In addition, the rigid nature of the probe should allow stability measures / recording, which is not possible with probes perfused catheters example.

We therefore propose to compare anal sphincter pressure in supine and standing, measured in high-resolution manometry.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over the age of 18 years
* Patient referred for endoscopic ultrasound and anal manometry anorectal HR-3D which is an indication of fecal incontinence or dyschesia

Exclusion Criteria:

* Patient age 18 Less
* Patient trust, guardianship, judicial protection
* No Written Consent
* Lack of social insurance
* History of anorectal surgery
* A presence of anal stenosis
* A setting evidence of anorectal lesion preventing the realization of the Screening
* Motor disability preventing the realization of the anorectal manometry 3D HR-standing situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
anal pressures measured by anorectal manometry and high-resolution three-dimensional | 12 months
  comparing two positions conventional position in the left lateral decubitus position with the feet.

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France